CLINICAL TRIAL: NCT03305848
Title: Efficacy and Safety of Oral Nitroglycerin on Esophageal Food Impaction
Brief Title: Esophageal Food Impaction
Acronym: ONEFIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A17-134
Record Dates: First submitted 2017-09-14; First posted 2017-10-10 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Food Bolus Obstruction
MeSH Terms: interventions — Nitroglycerin; Administration, Sublingual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oral nitroglycerin solution (Other): Up to 3 administrations of 0.4mg sublingual nitroglycerin tablets, dissolved in 10mL tap water, given orally in a single swallow. Each administration is separated by at least 5 minutes
  Interventions: Drug: Nitrostat 0.4Mg Sublingual Tablet

INTERVENTIONS:
Drug: Nitrostat 0.4Mg Sublingual Tablet — Up to 3 administrations of 0.4mg sublingual nitroglycerin tablets, dissolved in 10mL tap water, given orally in a single swallow. Each administration is separated by at least 5 minutes, and only if systolic blood pressure > 100 mmHg.

SUMMARY:
This study is designed to obtain data on the safety and efficacy of oral nitroglycerin solution for the treatment of esophageal food impaction in patients presenting to the Emergency Department with presumed esophageal food impaction. The main hypothesis is to determine the success rate of oral nitroglycerin solution in relieving the food impaction by assessing the resolution of symptoms and the ability of the patient to swallow.

DETAILED DESCRIPTION:
A piece of food stuck in the esophagus (the tube connecting the mouth to the stomach) is a relatively common occurrence, estimated at a rate of 13 episodes per 100,000 people per year, mostly men, and usually attributed to swallowed meat. The current standard of care for patients presenting to an Emergency Department with this problem includes a trial of medication, usually glucagon but sometimes a carbonated beverage, an injection of nitroglycerin, or benzodiazepines. The medical interventions mentioned above have not been shown to be significantly effective and have unwanted side effects; glucagon is known to cause nausea and vomiting and benzodiazepines can cause sedation and depressed breathing. If the medication fails to relieve the problem, the patient may require a procedure called endoscopy, where a video scope and retrieval tool are inserted into the esophagus to remove the piece of food. There is significant risk associated with endoscopy, including the risks of anesthesia as well as with the physical procedure itself. Endoscopy also results in a prolonged hospital stay due to the time required for the procedure, as well as from anesthesia recovery. The ideal treatment would be a safe, inexpensive, quickly effective medication without significant side effects that could be administered without sedation or extensive monitoring. Oral nitroglycerin solution might just be that intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Presentation consistent with esophageal food impaction
* Ability to swallow a small volume of liquid.

Exclusion Criteria:

* Intractable vomiting
* Hemodynamic instability or SBP <100 mmHg
* Concern for or evidence of significant airway compromise
* Concern for or evidence of esophageal perforation,
* Concern for or evidence of coronary ischemia
* Presentation > 12 hours since onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Stellpflug, MD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 patients were enrolled who met inclusion for the study.
Period: Overall Study
Arm/Group | Oral Nitroglycerin Solution
Started | 20
Completed | 17
Not Completed | 3
Not completed — Symptom resolution after consent, but before study drug administration | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: 17 of the 20 subjects received the study intervention.
Arm/Group | Oral Nitroglycerin Solution
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (19.08230098)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patients Condition at Discharge
Description: the proportion of study patients who achieve resolution of food impaction
Time Frame: Length of Emergency Department stay (Time Frame: up to 12 hours)]
Population: 17 of 20 enrolled subjects received the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Nitroglycerin Solution
Number analyzed (Participants) | 17
Participants
  Resolution with study treatment | 2
  Failure of resolution with study treatment | 15

2. Primary Outcome: Medications/Procedures Performed During Visit
Description: Total number of other medications or procedures used to relieve the esophageal food impaction
Time Frame: Length of Emergency Department stay (Time Frame: up to 12 hours)]
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Nitroglycerin Solution
Number analyzed (Participants) | 17
Participants
  Received additional medication | 7
  Underwent endoscopy | 15

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Oral Nitroglycerin Solution
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Nitroglycerin Solution (N=17)
Hypotension (Vascular disorders) | 1 (1) — SBP < 90
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03305848/Prot_SAP_000.pdf